CLINICAL TRIAL: NCT04794205
Title: Acute Changes In Thermal Pain Response Following Single Oral Dose of Beta-Cary
Acronym: BCP-Pain
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Delayed project onset; PI determined pilot data could be collected at a later date.
Sponsor: Hartford Hospital (Other)
Responsible Party: Principal Investigator, Godfrey Pearlson, Founding Director Olin Neuropsychiatry Research Center; Professor Yale University, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: HHC-2020-0365
Record Dates: First submitted 2021-03-03; First posted 2021-03-11 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Beta-Caryophyllene
Keywords: Beta-caryophyllene; Pain; BCP
MeSH Terms: conditions — Pain | interventions — caryophyllene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low Dose BCP (Experimental): Subjects will receive low dose of BCP.
  Interventions: Drug: Low Dose Beta-Caryophyllene
- Medium Dose BCP (Experimental): Subjects will receive a medium dose of BCP
  Interventions: Drug: Medium Dose Beta-Caryophyllene
- High Dose BCP (Experimental): Subjects will receive high dose of BCP.
  Interventions: Drug: High Dose Beta-Caryophyllene
- Placebo (Experimental): Subjects will receive placebo drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low Dose Beta-Caryophyllene — 5 mg BCP
  Other Names: Food grade BCP
  Arms: Low Dose BCP
Drug: Medium Dose Beta-Caryophyllene — 30 mg BCP
  Other Names: Food grade BCP
  Arms: Medium Dose BCP
Drug: High Dose Beta-Caryophyllene — 150 mg BCP
  Arms: High Dose BCP
Drug: Placebo — Placebo drug.
  Arms: Placebo

SUMMARY:
Beta-Caryophyllene is an essential oil and cannabis plant derivative also found in edible herbs. It has shown promise as a potential analgesic in preclinical trials. However, there are no human studies characterizing pharmacokinetics of BCP in humans. Therefore, it is of great importance to determine the pharmacokinetics of BCP in humans so that appropriate dosing can be developed for analgesia. This pharmacokinetic work will lay the groundwork for subsequent experiments testing the neural mechanism of BCP on pain.

DETAILED DESCRIPTION:
Chronic pain conditions are among the most common reasons adults seek medical care. Given the abuse potential for opioid analgesics, a substantial number of individuals with chronic pain have turned to alternatives such as medical marijuana. There is increasing evidence that medical marijuana has potential benefits for pain related conditions, but it also carries unwanted side effects such as impaired cognition and motor skills that may linger long after use, social stigma, and a moderate potential for abuse. Much of the marijuana/pain research is predicated on the assumption that its potential analgesic effects are due to its primary psychoactive ingredient - delta-9-tetrahydrocannabinol (THC). However, marijuana also contains dozens of phytochemicals, including cannabinoids and terpenes. Accordingly, there is interest in characterizing potential pain-relieving effects of these non-intoxicating constituents of marijuana. Thus far, it is unclear which components may be most relevant for influencing pain, or the mechanisms by which they exert their effects. Betacaryophyllene (BCP) may be a possible candidate because it is isolatable, has shown evidence as a potential analgesic in preclinical research, is known to be safe for human administration, and there is a strong premise for believing it interacts with the neurobiological systems in the brain that process pain.

This project was conceptualized to advance our mechanistic understanding of the analgesic potential of BCP in humans. The study will be a randomized, placebo-controlled, double-blind study of the pharmacokinetic mechanisms of BCP, including dosing and duration of action, and its potential analgesic effect on thermal pain induction following single-oral dosage. Ten healthy participants will be screened and on each of four subsequent visits will be dosed with either 5 mg, 30 mg, 150 mg of BCP or placebo. Participants' sensitivity to thermal pain induction will be measured before and after administration of the drug using a self survey of pain level. Successful completion of the project may elucidate the potential analgesic effects of ingesting beta-caryophyllene in humans, which can lead to new forms of treatment for pain.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of all races and ethnicities.
* 18/50 yrs old.
* Medically healthy (as determined by medical history and treatment).
* No current substance abuse disorder
* Adequate comprehension of English in order to complete study materials.
* Able and willing to provide written informed consent, and willing to commit to the study protocol.

Exclusion Criteria:

* Estimated premorbid intellectual disability <80 (WRAT-4)
* Neurological or medical disorder that may affect brain function.
* Comorbid DSM-V diagnosis of alcohol or substance abuse in prior 1 month or substance dependence in prior 3 months
* Vulnerable populations (e.g. pregnant, nursing, incarcerated); unwillingness to use reliable means of contraception.
* High risk for suicide defined as > 1 attempt in past 12 months that required medical attention, any attempt in the past 3 months or current suicidal ideation with plan and intent such that outpatient care is precluded.
* Current homicidal ideation with plan and intent such that outpatient care is precluded.
* Positive result on urine toxicology test for any substance, including CBD
* Any current acute or chronic pain condition
* Current use of any pain prescribed ROTC medications including opioids, NSAIDs, acetaminophen etc.
* Initial detection of abnormal liver function tests or CBC (see below)
* Initial detection of significant EKG abnormality

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Changes in self-rating for pain following ingestion of BCP. | Once immediately prior to drug administration; post drug administration at 1 and 2 hours.
  Participants will rate sensitivity to thermal pain induction using a visual analog scale post administration of BCP. The scale is titled "Thermal Pain Visual Analog Scale" and has values from 0 to 10 with 0 being the least painful and 10 being the most painful.

CONTACTS AND LOCATIONS:
Overall Officials: Godfrey Pearlson, MD, Principal Investigator — Founding Director Olin Research Center; Yale University
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided